CLINICAL TRIAL: NCT05091385
Title: The Efficacy of Mepolizumab in Patients With Severe Eosinophilic Asthma Treated in Poland. The Real-life Observational Study
Brief Title: Efficacy of Mepolizumab in Polish Patients With Severe Eosinophilic Asthma
Status: Completed | Type: Observational
Sponsor: Medical University of Lodz (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 10867
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-08

CONDITIONS: Asthma; Eosinophilic
Keywords: severe eosinophilic asthma; eosinophils; biological treatment; anti-interleukin(IL)-5; monoclonal antibody
MeSH Terms: conditions — Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Severe asthma patients treated with mepolizumab: Patients having received mepolizumab 100 mg SC every 4 weeks for at least 12 months in six severe-asthma clinics in Poland between December 2017 and December 2019
  Interventions: Biological: Mepolizumab given SC 100mg every 4 weeks between Dec 2017 and Dec 2019

INTERVENTIONS:
Biological: Mepolizumab given SC 100mg every 4 weeks between Dec 2017 and Dec 2019 — Mepolizumab administered within the frame of a severe asthma treatment program financed by National Health Fund in Poland for patients fulfilling specific criteria of asthma severity.

SUMMARY:
This study is aimed at evaluation of the efficacy of mepolizumab 100 mg subcutaneously (SC) every 4 weeks in patients with severe eosinophilic asthma who have been treated for at least 12 months in several Polish allergy/asthma centres under the same protocol. Target population to be recruited has been set at 130 subjects from at least 6 asthma centers throughout the country. Data on demographics and asthma status will be collected using questionnaires at 3 time-points: pre-mepolizumab (pre-MEPO), after 24 weeks of mepolizumab (MEPO) and after 1 year of MEPO administration (some of the outcomes will be observed every 4 weeks). Primary endpoints will include:

* Asthma exacerbations measured at qualification for the treatment (in the period of previous 52 weeks) and at the 24th and 52nd week of the treatment.
* Oral Corticosteroids use dose (documented at qualification for the treatment and at the 24th and 52nd week of the treatment).

DETAILED DESCRIPTION:
This study is aimed at evaluation of the efficacy of mepolizumab 100 mg SC every 4 weeks in patients with severe eosinophilic asthma who have been treated for at least 12 months in several Polish allergy/asthma centres under the same protocol. Retrospective multicentre observational study will involve 130 patients with severe eosinophilic asthma (SEA) who have been treated in six Severe Asthma Treatment Centres (SATCs) in Poland. In each SATC all data available in the program questionnaires will be transferred to the Study Data Sheet (questionnaire), and will be send to the study coordinator within 5 months from the study beginning The start-up meeting including partners from all centres involved will be organized to discuss the study protocol and to unify data collection The evaluation parameters (exacerbations rate, OCS dose) will be analysed at least at three time points: pre-MEPO, after 24 weeks of MEPO and after 1 year of MEPO administration (some of the outcomes will be observed every 4 weeks, for the details see 'study endpoints' section).

In addition the following parameters which are available in patients' records will be analysed:

* 5-item asthma control questionnaire (ACQ-5) score (measured at qualification for the treatment and every 4 weeks thereafter)
* Asthma quality of life questionnaire (AQLQ) score (measured at qualification for the treatment and every 4 weeks thereafter)
* Pre-bronchodilator FEV1 (measured at qualification for the treatment and every 4 weeks thereafter)

Research activities will include:

* collecting raw data from the clinical centres (paper version) and constructing a raw dataset (digital version),
* data cleaning, computation of variables,
* statistical analysis typical for pre-post study design (the statistical analysis will be outsourced to the specialized private institute).

Clinical improvements observed at 24 weeks and at 52 weeks of treatment with Mepolizumab will be referred to the following characteristics of patients at baseline:

* demographics,
* presence of comorbidities including the atopic status,
* concomitant pharmacotherapy,
* clinical status,
* eosinophilia. We will control for mepolizumab use regarding dose, treatment duration and dosing frequency as well as for the safety profile based on the AEs reporting in the medical documentation.

Data Source / Data Collection Patients recruited to the study had been treated with mepolizumab between December 2017 and December 2019.All the data planned to be used in the proposed study were systematically collected in the form of the clinical documentation (paper version) and will be transferred in the study centres into the study.

Data Sheets. Collaborating Researchers (Severe Asthma Centres' Leaders) will provide the data input into the dedicated online questionnaire.

Study Population 130 Patients who were treated with mepolizumab in six severe-asthma clinics in Poland between December 2017 and December 2019 . In the drug program in Poland it was mandatory to conduct the control examinations at the 24th and 52nd week of the treatment . In the proposed study we will use this information to evaluate study endpoints. Only patients who have been treated for at least 52 weeks are included into the study

Variables concerning the primary endpoints

* Asthma exacerbations measured at qualification for the treatment (in the period of previous 52 weeks) and at the 24th and 52nd week of the treatment.
* Oral Corticosteroids use dose (documented at qualification for the treatment and at the 24th and 52nd week of the treatment)

Variables concerning the secondary endpoints:

* ACQ-5 score (measured at qualification for the treatment and every 4 weeks thereafter)
* AQLQ score (measured at qualification for the treatment and every 4 weeks thereafter)
* Pre-bronchodilator forced expiratory volume in 1 second (FEV1) (measured at qualification for the treatment and every 4 weeks thereafter)
* Blood eosinophil counts (measured at qualification for the treatment and at the 24th and 52nd week of the treatment)

ELIGIBILITY:
Inclusion Criteria:

* The availability of the complete data

* Duration of treatment with mepolizumab: ≥ 52 weeks
* Satisfying the Polish drug programme inclusion criteria:
* Age >18
* Before treatment with mepolizumab (BSAT inclusion criteria):

  * High doses of inhaled corticosteroids (ICS) + one other controlling medication (i.e. LABA)
  * ≥2 exacerbations in the previous year
  * ≥350 eosinophil cells/microliter (µl) in the peripheral blood at the time of qualification or in the previous year
  * Pre-bronchodilator FEV1 < 80%

Exclusion Criteria:

* Duration of treatment with mepolizumab < 52 weeks

• Lack of complete data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 130 Patients who were treated with mepolizumab in six severe-asthma clinics in Poland between December 2017 and December 2019 . In the drug program in Poland it was mandatory to conduct the control examinations at the 24th and 52nd week of treatment. In the proposed study we will use this information to evaluate study endpoints. Only patients who have been treated for at least 52 weeks are included into the study.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Kurowski, MD, PhD, Principal Investigator — Medical University of Lodz
Locations (1):
- Medical University of Lodz, Dept. of Immunology and Allergy, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Yes
Individual entries regarding laboratory results, concomitant medications, comorbidities and clinical features of asthma exacerbations will be made available upon request, as specified below.
Supporting Information: CSR
Access Criteria: The data may be received upon reasonable written request form the principal investigator.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients having received mepolizumab 100 mg SC every 4 weeks for at least 12 months in six severe-asthma clinics in Poland between December 2017 and December 2019
Pre-assignment Details: Not applicable. A uniform, single treatment group throughout the study. No wash-out or run-in periods.
Period: Overall Study
Arm/Group | Severe Asthma Patients Treated With Mepolizumab
Started | 106
Completed | 106
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Group: Patients having received mepolizumab 100 mg SC every 4 weeks for at least 12 months in six severe-asthma clinics in Poland between December 2017 and December 2019
Arm/Group | Study Group
Number analyzed (Participants) | 106
Age, Customized [Median (Inter-Quartile Range); unit: years] — Age criterion for recruitment was 18 years or older at the time of treatment initiation. Population: Initially 130 subjects had been recruited, of whom complete data for 106 had been collected, and those subjects were included into the analysis.
  years
    Age | 56.6 [49 to 66]
Sex: Female, Male [Count of Participants; unit: Participants] — 77 out of 106 analyzed subjects were females (72.6%) Population: 106 subjects with complete data were finally analyzed
  Participants
    Female | 77
    Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Patients were recruited in six severe asthma centers in Poland
  Participants
    Poland | 106

OUTCOME MEASURES:

1. Primary Outcome: Asthma Exacerbations During 52 Weeks Preceding Treatment Initiation (as Assessed at Baseline) and at the 24th and 52nd Week of the Treatment
Description: Data as transferred from the treatment program questionnaires to the Study Data Sheet. Asthma exacerbations, defined according to the Polish drug programme, is the worsening in asthma requiring (1) use of systemic corticosteroids or (2) increase in dose of OCS for more than 3 days in case of patients who are chronically treated with OCS.
Time Frame: Baseline (before mepolizumab initiation); week 24; week 52
Measure: Median (Inter-Quartile Range); unit: number of asthma exacerbations
Arm/Group | Study Group
Number analyzed (Participants) | 106
number of asthma exacerbations
  baseline exacerbations number | 3 [2 to 5]
  Exacerbations at week 24 | 0 [0 to 1]
  Exacerbations at week 52 | 0 [0 to 1]

2. Primary Outcome: Number Patients Requiring Treatment With Oral Corticosteroids (OCS) at a Chronic Basis (Documented at Qualification for the Treatment and at the 24th and 52nd Week of the Treatment)
Description: Data as transferred from the treatment program questionnaires to the Study Data Sheet
Time Frame: Baseline (before mepolizumab initiation); week 24; week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 106
Participants
  Participants requiring chronic OCS treatment of asthma BASELINE | 70
  Participants requiring chronic OCS treatment of asthma week 24 | 20
  Participants requiring chronic OCS treatment of asthma week 52 | 15

3. Secondary Outcome: ACQ-5 (Asthma Control Questionnaire 5-item) Score
Description: Asthma Control Questionnaire (ACQ) is the validated tool aimed to measure the adequacy of asthma control and change in asthma control occurring either spontaneously or as a result of treatment. It is self-administered by patients and assesses asthma symptoms intensity and frequency (5 items) on a 7-point scale (0 through 6; 0=absence, 6= maximum intensity/frequency), with total score being the average of the questions. ACQ score ranges from 0 (minimum) to 6 (maximum). A score of 1.5 or more indicates that a patient has inadequate asthma control. Difference in score of 0.5 or greater is considered clinically important (MCID, minimal clinically important difference).
Time Frame: Baseline (before mepolizumab initiation); week 24; week 52
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 106
scores on a scale
  ACQ score value BASELINE | 3.48 [2.82 to 4.45]
  ACQ score value week 24 | 1.53 [0.80 to 2.47]
  ACQ score value week 52 | 1.31 [0.66 to 2.12]

4. Secondary Outcome: AQLQ (Asthma Quality of Life Questionnaire) Score
Description: Asthma Quality of Life Questionnaire (AQLQ) is a disease-specific tool covering both physical and emotional impact of asthma upon the affected subjects' quality of life. This questionnaire has 4 domains: symptoms, activity limitation, emotional function, and environmental stimuli. The AQLQ has been validated in 2 variants: a standard AQLQ consisting of 32 items and a mini-AQLQ containing 15 items. In the national severe asthma treatment program in Poland a 15-item AQLQ is used, as per National Health Fund requirements. Items are scored on a 7-point Likert scale, with score 1 representing maximal impairment and the value of 7 attributed to "no impairment". The total score is calculated as a mean value of all items (a sum of scores divided by 15). A change of >0.5 points is considered clinically significant. Score below 5 indicates considerable lowering of quality of life in an asthmatic subject and is one of the conditions for inclusion into the reimbursed treatment program.
Time Frame: Baseline (before mepolizumab initiation); week 24; week 52
Measure: Median (Inter-Quartile Range); unit: score points
Arm/Group | Study Group
Number analyzed (Participants) | 106
score points
  AQLQ score BASELINE | 2.47 [1.19 to 3.50]
  AQLQ score week 24 | 5.8 [4.2 to 6.7]
  AQLQ score week 52 | 5.3 [4.25 to 6.3]

5. Secondary Outcome: Pre-bronchodilator FEV1
Description: Pre-bronchodilator FEV1 (forced expiratory volume in 1 second) is a key indicator in lung funtion testing, measuring the volume of air exhaled from the lungs in the first second of a maximum forced exhalation. FEV1 is commonly used to diagnose and monitor obstructive lung diseases, including asthma. Values below 80% of the predicted value (calculated individually using basing on subject's age, sex, height, weight and ethnicity) indicates narrowing of the airways.
Time Frame: Baseline (before mepolizumab initiation); week 24; week 52
Measure: Median (Inter-Quartile Range); unit: % predicted
Arm/Group | Study Group
Number analyzed (Participants) | 106
% predicted
  FEV1 Baseline | 62 [50 to 75]
  FEV1 week 24 | 76.0 [60.3 to 85.7]
  FEV1 week 52 | 76 [62 to 85.2]

6. Secondary Outcome: Blood Eosinophil Counts
Description: Data as transferred from the treatment program questionnaires to the Study Data Sheet
Time Frame: Baseline (before mepolizumab initiation); week 24; week 52
Measure: Median (Inter-Quartile Range); unit: cell per microliter
Arm/Group | Study Group
Number analyzed (Participants) | 106
cell per microliter
  Eosinophil count (peripheral blood) BASELINE | 605 [430 to 800]
  Eosinophil count (peripheral blood) week 24 | 60 [30 to 100]
  Eosinophil count (peripheral blood) week 52 | 60 [30 to 110]

ADVERSE EVENTS:
Time Frame: Throughout the treatment period (weeks 0 through 52)
Description: Two (1.9%) patients were reported to experience adverse events during treatment. One (0.9%) patient experienced a miscarriage after 7th dose of mepolizumab administration. One (0.9%) patient complained of pain in the small joints of the both hands
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 2/106
Serious Adverse Events (participants affected / at risk) | 1/106
Other Adverse Events (participants affected / at risk) | 1/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=106)
miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 (1) — occurred after 7th dose, other details not reported
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=106)
pain in the small joints of both hands (Musculoskeletal and connective tissue disorders) | 1 (1) — no more details known, mild and transient

LIMITATIONS AND CAVEATS:
Retrospective study, basing on reports from national health data system (as per requirements of national health insurance fund). Incompleteness of data for 24 patients, not possible to be retrieved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT05091385/Prot_SAP_000.pdf